CLINICAL TRIAL: NCT06248489
Title: Examination of Manual Skills in Individuals With and Without Chronic Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU_Erol_10
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with neck pain
- Individuals without neck pain

SUMMARY:
This study will determine whether manual dexterity is affected in individuals with neck pain compared to individuals without neck pain. It is thought that determining the changes in dexterity in individuals with neck pain compared to healthy individuals will shed light on future more detailed studies on the current subject.

ELIGIBILITY:
Inclusion Criteria:

- Experiencing neck pain for at least 3 months

Exclusion Criteria:

- Having another medical condition that may affect dexterity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neck pain
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline
  While the left end of a 10 cm line represents no pain, the right end represents unbearable pain.
9 hole peg test | Baseline
  It is a brief, standardized, quantitative upper extremity function test that measures manual dexterity.
The Bournemouth Questionnaire for Neck Pain | Baseline
  It consists of 7 questions examining pain intensity, activities of daily living, social activities, anxiety, emotional aspects of depression, kinesiophobia, and the ability to control pain.
The Fremantle Neck Awareness Questionnaire | Baseline
  It is a 9-question survey that evaluates neck perception, attention and proprioceptive awareness in individuals with neck pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)